CLINICAL TRIAL: NCT06926855
Title: Community Health Workers Systematically Assessing and Addressing Social Determinants of Health to Improve Outcomes in Community Health Centers (CHW-SYSTIM)
Brief Title: Community Health Workers Reduce Social Barriers That Affect the Health of Patients With High Blood Pressure and Diabetes.
Acronym: (CHW-SYSTIM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Health Choice Network (Other); OCHIN, Inc. (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Westat (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2168673-4; NHLBI Sub-Other Transaction (Other: National Institutes of Health(NIH)/National Heart, Lung and Blood Institute(NHLBI))
Record Dates: First submitted 2025-02-28; First posted 2025-04-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Uncontrolled Diabetes; Uncontrolled Hypertension
Keywords: Uncontrolled diabetes; Federally Qualified Health Center (FQHC); Community Health Worker (CHW); CEAL; Randomized Controlled Trial (RCT); Social Determinants of Health (SDOH); Social Needs; Diabetes Mellitus; Hemoglobin A1C; Advanced Encryption Standard; Uncontrolled hypertension; health differences
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Community Health Centers (Experimental): Community Health Centers (CHC) will identify a Community Health Worker (CHW) or similar staff member who will conduct social risk activities as part of clinical services for all CHC patients with uncontrolled diabetes (DM) and hypertension (HTN) as defined by Uniform Data System (UDS). If needed due to resource constraints, a prioritization scheme may be applied to target patients with the most poorly controlled DM / HTN, those newly diagnosed, those at selected CHC-run sites, etc.; this scheme will be refined in the intervention development phase.
  Interventions: Other: CHC-level cluster randomized control trial
- Control Community Health Centers (No Intervention): Control CHC data on enabling services and associated workflows will be gathered through qualitative methods for a deeper understanding of the intervention impact. At the end of the intervention year, control CHCs will receive: (1) participation in the end of intervention summative CHW convening for crossover training led by the intervention arm CHWs; and 2) a toolkit designed to support their adoption of the intervention processes. This will both support the dissemination of intervention elements identified as effective (as feasible), and recruitment activities (by ensuring that all study FQHCs receive something through study participation).

INTERVENTIONS:
Other: CHC-level cluster randomized control trial — CHW (with clinic champion support) outreach to eligible patients, verbally consent patients, confirm eligibility, conduct social needs screening, make service or resource referrals, plan and support referral completion as needed, follow-up with patients to assess referral completion and outcomes
  Implementation supports: financial support for CHW, clinic champion, and CHC administration of trial activities; 12 weeks of preparatory CHW training and coaching; practice coaching and technical support for data collection at all sites; additional support for sites without existing research data infrastructure; CHW Learning Collaborative through intervention and follow-up period for implementation support and cross-training control sites.
  Arms: Intervention Community Health Centers

SUMMARY:
The goal of this mixed-methods study is to assess the impact of a Community Health Worker (CHW)-led social risk screening and referral in improving management of uncontrolled diabetes (DM) and hypertension (HTN) among patients receiving care in community health centers (CHCs or health centers). The intervention is focused on adult health center patients with uncontrolled DM and/or HTN. Study findings will provide important evidence to guide CHCs in implementing programs to address social risks in their patient populations. Findings will illuminate whether and how CHW-led interventions to address social needs yield the hypothesized outcomes. The aims of the study are:

* AIM 1: Measure how effective the CHW-led social risk program is at reducing blood sugar levels (A1C) in CHC patients with uncontrolled DM and lowering blood pressure in CHC patients with uncontrolled HTN.
* AIM 2: Identify effective strategies for increasing and expanding CHW-led social risk programs.

DETAILED DESCRIPTION:
BACKGROUND: Social determinants of health (SDOH) are the conditions of the environment in which people are born, live, work, and age; they are non-medical factors that impact health. Adverse SDOH are often called social risks; when patients report having such risks and desiring strategies for mitigating them, it is often called social needs. Exposure to social risks contributes to numerous poor health outcomes and is associated with negative impacts on chronic disease outcomes like diabetes (DM) and hypertension (HTN) control.

People with HTN have high rates of social risks, and these rates are higher among African American, Alaskan Native, American Indian, Native Hawaiian and Pacific Islander patients than white patients. Social risks often occur in clusters, and patients with multiple social risks are more likely to have uncontrolled DM and / or uncontrolled HTN. Given the many negative health impacts of social risks, numerous national guidelines recommend screening for and addressing social risks through referral to social services. The impacts of social risks on DM and HTN outcomes are most profound in the communities served by community health centers (CHCs). CHC patients with DM have high rates of unmet social needs. Therefore, the need for interventions that mitigate the impacts of social risks on these chronic disease outcomes - and the need for evidence on how to implement such interventions effectively and sustainably - is critical in the CHC setting.

Many CHCs strive to assess and address social risks but lack an approach to doing so systematically; as a result, not all patients who could benefit from such efforts - such as those with uncontrolled DM and / or HTN - do so. The many known barriers to widespread adoption of systematic social risk screening and referral-making include challenges associated with fitting social risk screening, documentation, and referral-making into clinic workflows.

Preliminary evidence suggests that Community Health Workers (CHWs) could play a critical part in CHC approaches to identifying social risks and referring patients with social needs to social services. CHW models of care have been shown to have a significant and positive impact on health outcomes, including hospitalization readmission rates and continuity of care. Thus, CHW-based approaches in CHCs might mitigate the impacts of social risks on DM and HTN. However, given the substantial barriers to implementing social risk-related activities in clinical settings, research is needed on how to optimize CHW-focused social risk interventions, and how to implement such interventions so they are adopted systematically and sustainably. Yet there are barriers specific to CHWs' potential ability to support CHCs' social risk efforts, including CHWs' large caseloads, competing demands, and time pressure, limited ability to enter data in the electronic health record, and CHWs lacking needed information to connect patients with social services. Thus, there is a clear need for research on: the impact on DM and HTN outcomes of CHW-led interventions to address social risks, whether and how CHW-led interventions support implementing this model in CHCs, and strategies for enhancing the sustained implementation of CHW-led interventions in this setting. The proposed study will generate some of this needed evidence.

SETTING: The RCT will be conducted in CHCs. NCPCR, comprised of two research networks (OCHIN, Morehouse School of Medicine (MSM)), will engage three primary care networks (OCHIN, Health Choice Network (HCN), and the Southeast Regional Clinicians Network (SERCN)) and these existing networks will be leveraged to recruit CHCs to participate in the RCT.

STUDY POPULATION: Adult patients ≥18 years old receiving care in one of the participating CHCs, with a DM diagnosis and most recent A1c >9, and / or a HTN diagnosis and last systolic BP >140 or last diastolic BP >90.

DATA COLLECTION:

1. Electronic Health Record (EHR) data: The study will obtain de-identified EHR data from CHCs for patients ages 18 years and older. This data has already been collected as part of regular patient care. All data will be de-identified, so there is minimal risk of identification. EHR data will also be de-identified, and it is not practical to attain consent for the utilization of EHR data. The data will include patient demographics, health center characteristics, SDOH data, and clinical outcomes (i.e., % targeted patients with improved BP, % targeted patients with improved HbA1c, % targeted patients with new BP measures documented every >=3 months after first CHW contact, % targeted patients with DM with new HbA1c measures documented every >=3 months after first CHW contact).
2. CHW-collected REDCap data (Intervention sites): The study will also collect common prospective data elements to assess the delivery of the intervention. This data will be collected in a separate data management system (i.e., REDCap) by the CHWs. The data will include % targeted patients with up-to-date SDOH screening by end of follow-up period, % patients with social risks that received a referral, % of patients with patient self-reported receipt of the recommended services. The no Intervention CHCs will receive access to standard online CHW training modules free of charge to them.
3. Qualitative data: The study team will conduct 1) virtual semi-structured interviews with a subset of the CHW staff to explore their experiences, perspectives, successes, and challenges; 2) CHC-specific virtual group interviews will focus on context/setting and referral processes; hopes, expectations and perceived challenges regarding the intervention; perceived impact of the intervention on social risk screening and referral; patient care access and quality (including any negative impacts); clinical workflow and staff reactions/satisfaction; expectations met or unmet and challenges encountered during the intervention; and lessons learned; and 3) cross-CHC virtual patient focus groups or interviews to explore patient experience with and reactions to the CHW-led screening and referral process, including any impact (positive or negative) on their perception of the care they received, their relationships with members of the care team, their ability to access material support, and their health.

In this concurrent mixed methods study, quantitative and qualitative data are collected in parallel and initially analyzed separately. Once preliminary analyses are complete, quantitative and qualitative analysts will meet to share results and work to integrate the mixed method data and present the combined data, organized by RE-AIM domain.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* People with Type 2 diabetes with their most recent hemoglobin A1c test result (a blood test that reflects average blood sugar levels over the past 2-3 months) is greater than or equal to 9%.
* People with essential hypertension with their last systolic blood pressure (BP) (the top number in a BP reading) is greater than or equal to 140 mmHg or diastolic BP (the bottom number in a BP reading) is greater than or equal to 90 mmHg.

Exclusion Criteria

* People who are less than 18 years old
* Pregnant people
* People who don't meet the Type 2 diabetes or hypertension criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Test the hypothesis that CHW-led process will improve health outcomes among DM patients post 12 month intervention | Measured at 6 months and 12 months after the first CHW contact.
  Percentage of participants with any reduction in HgbA1C from baseline.
Test the hypothesis that CHW-led process will improve health outcomes among HTN patients post 12 month intervention | Measured at 6 months and 12 months after the first CHW contact.
  Percentage of participants with any reduction in systolic and/or diastolic blood pressure from baseline.

SECONDARY OUTCOMES:
Assess the provision of appropriate social need screening | Social needs screening conducted during the 6 months intervention period.
  Percentage of CHC patients who received social needs screening from the CHW.
Assess percentage of patients referred to social services | Referral assessed at 6 months after first CHW contact.
  Percentage of CHC patients were referred to social services.
Assessing successful patient service linkage rate | Successful linkage assessed at 12 months after first CHW contact.
  Percentage of CHC patients who were successfully linked to services.
Evaluating Staff Experiences through Interviews and Surveys on Implementation Strategies | Assessed at study completion (up to 12 months after the first CHW contact)
  Qualitative assessment of CHW and CHC staff experiences with implementation strategies through staff interviews and surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Douglas, JD, Principal Investigator — Morehouse School of Medicine; Rachel Gold, PhD, MPH, Principal Investigator — OCHIN, Inc.; Katherine Chung-Bridges, MD, MPH, Principal Investigator — Health Choice Network (HCN)
Locations (3):
- United States (3):
  - Health Choice Network (HCN), Miami, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - OCHIN, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
In alignment with NIH data sharing policies and organizational agreements, we will develop a process for sharing RCT data once the study is complete. RCT data will be available as follows:
  For patients in the RCT intervention sites who provide informed consent, de-identified patient-level data will be available for future research, per NIH's DMSP. In alignment with NIH data sharing policies and organizational agreements, we will develop a process for sharing RCT data once the study is complete.
  For patients who are not consented (i.e. ALL patients in control clinics and any patients in intervention clinics who are not consented), only aggregate data can be shared. Aggregate data are defined as a dataset or data display that consolidates data from multiple individuals (e.g., patients) and does not contain identifiers that can be used to identify individual patients.
Supporting Information: Study Protocol, CSR
Time Frame: July 1st, 2026 - June 30th, 2028

REFERENCES:
- [Background] Ruiz Escobar E, Pathak S, Blanchard CM. Screening and Referral Care Delivery Services and Unmet Health-Related Social Needs: A Systematic Review. Prev Chronic Dis. 2021 Aug 12;18:E78. doi: 10.5888/pcd18.200569. PMID 34387188
- [Background] Carter J, Hassan S, Walton A, Yu L, Donelan K, Thorndike AN. Effect of Community Health Workers on 30-Day Hospital Readmissions in an Accountable Care Organization Population: A Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e2110936. doi: 10.1001/jamanetworkopen.2021.10936. PMID 34014324
- [Background] Greenwood-Ericksen M, DeJonckheere M, Syed F, Choudhury N, Cohen AJ, Tipirneni R. Implementation of Health-Related Social Needs Screening at Michigan Health Centers: A Qualitative Study. Ann Fam Med. 2021 Jul-Aug;19(4):310-317. doi: 10.1370/afm.2690. PMID 34264836
- [Background] Cockerham WC, Hamby BW, Oates GR. The Social Determinants of Chronic Disease. Am J Prev Med. 2017 Jan;52(1S1):S5-S12. doi: 10.1016/j.amepre.2016.09.010. PMID 27989293
- [Background] Balfour PC Jr, Rodriguez CJ, Ferdinand KC. The Role of Hypertension in Race-Ethnic Disparities in Cardiovascular Disease. Curr Cardiovasc Risk Rep. 2015 Apr;9(4):18. doi: 10.1007/s12170-015-0446-5. PMID 26401192
- [Background] Yan AF, Chen Z, Wang Y, Campbell JA, Xue QL, Williams MY, Weinhardt LS, Egede LE. Effectiveness of Social Needs Screening and Interventions in Clinical Settings on Utilization, Cost, and Clinical Outcomes: A Systematic Review. Health Equity. 2022 Jun 24;6(1):454-475. doi: 10.1089/heq.2022.0010. eCollection 2022. PMID 35801145
- [Background] Krieger J, Collier C, Song L, Martin D. Linking community-based blood pressure measurement to clinical care: a randomized controlled trial of outreach and tracking by community health workers. Am J Public Health. 1999 Jun;89(6):856-61. doi: 10.2105/ajph.89.6.856. PMID 10358675
- [Background] Kangovi S, Mitra N, Norton L, Harte R, Zhao X, Carter T, Grande D, Long JA. Effect of Community Health Worker Support on Clinical Outcomes of Low-Income Patients Across Primary Care Facilities: A Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1635-1643. doi: 10.1001/jamainternmed.2018.4630. PMID 30422224
- [Background] Hartzler AL, Tuzzio L, Hsu C, Wagner EH. Roles and Functions of Community Health Workers in Primary Care. Ann Fam Med. 2018 May;16(3):240-245. doi: 10.1370/afm.2208. PMID 29760028
- [Background] Sandhu S, Lian T, Smeltz L, Drake C, Eisenson H, Bettger JP. Patient Barriers to Accessing Referred Resources for Unmet Social Needs. J Am Board Fam Med. 2022 Jul-Aug;35(4):793-802. doi: 10.3122/jabfm.2022.04.210462. PMID 35896446
- [Background] Browne J, Mccurley JL, Fung V, Levy DE, Clark CR, Thorndike AN. Addressing Social Determinants of Health Identified by Systematic Screening in a Medicaid Accountable Care Organization: A Qualitative Study. J Prim Care Community Health. 2021 Jan-Dec;12:2150132721993651. doi: 10.1177/2150132721993651. PMID 33576286
- [Background] Wan W, Li V, Chin MH, Faldmo DN, Hoefling E, Proser M, Weir RC. Development of PRAPARE Social Determinants of Health Clusters and Correlation with Diabetes and Hypertension Outcomes. J Am Board Fam Med. 2022 Jul-Aug;35(4):668-679. doi: 10.3122/jabfm.2022.04.200462. PMID 35896473
- [Background] Daly A, Sapra A, Albers CE, Dufner AM, Bhandari P. Food Insecurity and Diabetes: The Role of Federally Qualified Health Centers as Pillars of Community Health. Cureus. 2021 Mar 12;13(3):e13841. doi: 10.7759/cureus.13841. PMID 33854855
- [Background] Milani RV, Price-Haywood EG, Burton JH, Wilt J, Entwisle J, Lavie CJ. Racial Differences and Social Determinants of Health in Achieving Hypertension Control. Mayo Clin Proc. 2022 Aug;97(8):1462-1471. doi: 10.1016/j.mayocp.2022.01.035. Epub 2022 Jul 19. PMID 35868877
- See also: Centers for Disease Control and Prevention. (2030). Healthy People. — https://health.gov/healthypeople/priority-areas/social-determinants-health
- See also: Community health center chartbook 2023. — https://www.nachc.org/resource/community-health-center-chartbook-2022/.
- See also: National Academies of Sciences, Engineering, and Medicine. Investing in interventions that address non-medical, health-related social needs: Proceedings of a workshop. — https://nap.nationalacademies.org/catalog/25544/investing-in-interventions-that-address-non-medical-health-related-social-needs
- See also: Building the evidence base for social determinants of health interventions — https://aspe.hhs.gov/reports/building-evidence-base-social-determinants-health-interventions